CLINICAL TRIAL: NCT03792399
Title: Impact of Innovative Technology on Geriatric Diabetic Patients: Evaluation of Quality of Life, Self Efficacy and Glycemic Control Among Patients With Experience of Continuous Glucose Monitoring
Brief Title: Continuous Glucose Monitoring With Immediate or Delayed Counseling Feedback
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NCKUH-10508011
Record Dates: First submitted 2018-11-08; First posted 2019-01-03 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2018-11

CONDITIONS: Type2 Diabetes
Keywords: continuous glucose monitoring; immediate feedback counseling; delayed feedback counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate feedback counseling (Experimental): Professional CGM calibrate blood glucose via a glucsoe-oxidase-impregnated membrane during a 5 day period. The patient wearing professional CGM is randomized to immediate feedback after data downloaded into computer.
  Interventions: Behavioral: feedback counseling
- Delayed feedback counseling (Other): Professional CGM calibrate blood glucose via a glucsoe-oxidase-impregnated membrane during a 5 day period. The patient wearing professional CGM is randomized to delayed feedback (standard care, i.e., CGM graphs interpretation at scheduled 3 months outpatient visit).
  Interventions: Behavioral: feedback counseling

INTERVENTIONS:
Behavioral: feedback counseling — Professoinal CGM in combination with diet and exercise record is used as teaching material to help patient realize their blood glucose pattern and to modify their behavior after counseling feedback.

SUMMARY:
This study is designed to explore the effect of feedback counseling using professional continuous glucose monitoring on glycemic control, self-efficacy, and self-management behaviors among middle aged and older adults with poor controlled type 2 diabetes mellitus. This study also explores the difference on timing of feedback after continuous glucose monitoring exam.

DETAILED DESCRIPTION:
After scheduled routine professional continuous glucose monitoring (CGM) exam, participants in both the intervention and control group receive ordinary education and regimen adjustment as indicated based on CGM results. For participants in the intervention group, they will also receive CGM counseling immediately on the day of CGM sensor removal. For participants in the control group, they will receive CGM counseling on the day of routine 3 months outpatient visit.

Qualitative data are collected through in-depth interview: User expectation, acceptability and satisfaction of CGM are also explored during in-depth interview with a semi-structured questionnaire.

Quantitative data were collected through validated questionnaires, including evaluation of depression by a short form of the Center for Epidemiologic Studies Depression Scale Revised (CES-D-R), emotional stress by Problem Areas in Diabetes Scale (PAID), self efficacy by Stanford Self-Efficacy for Diabetes (SES), at pretest and 3 months after CGM counseling.

Anthropometric Measurements. Body height, body weight, body mass index, and blood pressure were recorded at pre-test and post-test interview.

Blood Tests. Routine biochemistry, fasting plasma glucose, hemoglobin A1c (HbA1c) are collected within 2 weeks of pretest and posttest day.

ELIGIBILITY:
Inclusion Criteria:

* Age 45 years old or more at recent outpatient visits;
* Type 2 diabetic patients followed up at National Cheng Kung University Hospital;
* Patients planned to receive CGM suggested by primary care physician due to inadequate controlled blood glucose.

Exclusion Criteria:

* Patients with diagnosis of generalized inflammation, advanced malignancy, end-stage renal disease on regular dialysis, status post renal transplantation, end-stage liver, heart or pulmonary disease;
* Patients who are taking systemic glucocorticoids;
* Any acute or chronic inflammatory disease as determined by a leukocyte count over 10,000/mm3 or clinical signs of infection;
* Patients who could not complete the questionnaires or who could not follow order due to cognitive impairment or in bed-ridden status;
* Patients diagnosed as thalassemia, glucose-6-phosphate dehydrogenase deficiency, and any other hemoglobinopathies that may influence the accuracy of hemoglobulin A1c measurement were also excluded. Patients who received blood transfusion in recent 3 months were also excluded.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-03-07 (Actual); Primary Completion 2017-10-12 (Actual); Study Completion 2017-10-12 (Actual)

PRIMARY OUTCOMES:
Change of HbA1c | Baseline and 3 months after CGM counseling
  Change of HbA1c in 3 months after CGM counseling.
Change of score for self efficacy | Baseline and 3 months after CGM counseling
  Change of Stanford Self-Efficacy for Diabetes Scale (SES) in 3 months after CGM counseling. The score for each item ranged from 1-10. The score of the scale is the mean of the eight items. Higher number indicated higher self-efficacy.

SECONDARY OUTCOMES:
Change of score for diabetes associated stress | Baseline and 3 months after CGM counseling
  Change of score for Problem Areas in Diabetes Scale (PAID) in 3 months after CGM counseling. PAID is a 20-item self-reported questionnaire with scale 0-4 for each question, generating a total score of 0-100. A score of ≥ 40 is defined as emotional burnout.
Change of score for depression | Baseline and 3 months after CGM counseling
  Change of score for Center for Epidemiologic Studies Depression Scale Revised (CESD-R) in 3 months after CGM counseling. With 10-ietm CESD-R scale scoring 10 or more defined as having depression (range 0 to 30).
Change in diet composition | Baseline and 3 months after CGM counseling
  Change of carbohydrate amounts, fruits amount in 3 months after CGM counseling.
Change in exercise amount, time spent in light activity | Baseline and 3 months after CGM counseling
  Exercise amount recorded by acelerometers, built in sports bracelet (Fitbit Charge HRTM Wireless Heart Rate + Activity Wristband). Time spent in light activity per day in 3 months after CGM counseling feedback is compared with baseline.
Change in exercise amount, time spent in moderate activity | Baseline and 3 months after CGM counseling
  Exercise amount recorded by acelerometers, built in sports bracelet (Fitbit Charge HRTM Wireless Heart Rate + Activity Wristband). Time spent in moderate activity per day in 3 months after CGM counseling feedback is compared with baseline.
Change in exercise amount, time spent in intense activity | Baseline and 3 months after CGM counseling
  Exercise amount recorded by acelerometers, built in sports bracelet (Fitbit Charge HRTM Wireless Heart Rate + Activity Wristband). Time spent in intense activity per day in 3 months after CGM counseling feedback is compared with baseline.
Change in exercise amount (time spent in sedentary behavior) | Baseline and 3 months after CGM counseling
  Exercise amount recorded by acelerometers, built in sports bracelet (Fitbit Charge HRTM Wireless Heart Rate + Activity Wristband). Time spent in sedentary behavior in 3 months after CGM counseling feedback is compared with baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Ju Chiu, Ph.D., Study Director — Institute of Gerontology, NCKU; Ye-Fong Du, M.D., Principal Investigator — NCKUH

IPD SHARING:
Plan to Share IPD: Undecided
The study protocol will be shared after study publication.

REFERENCES:
- [Background] Allen NA, Fain JA, Braun B, Chipkin SR. Continuous glucose monitoring counseling improves physical activity behaviors of individuals with type 2 diabetes: A randomized clinical trial. Diabetes Res Clin Pract. 2008 Jun;80(3):371-9. doi: 10.1016/j.diabres.2008.01.006. Epub 2008 Mar 4. PMID 18304674